CLINICAL TRIAL: NCT02556775
Title: Pregnancy Registry to Collect Long-Term Safety Data From Women Treated With HyQvia
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 161301; EUPAS5798 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2015-06-26; First posted 2015-09-22 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Exposure During Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 33 Months
Biospecimen Retention: Samples Without DNA — Blood samples (plasma) for anti-recombinant human hyaluronidase (rHuPH20) antibodies that remain after study testing is done may be stored and used for additional testing (eg, further evaluation of an abnormal test or an adverse event). Samples will be stored in a coded form for a maximum of 2 years after the final study report has been completed and, subsequently, will be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alternative Product Arm: Participant stops HYQVIA treatment (if the participant is still treated) and a licensed human normal immunoglobulin other than HYQVIA for intravenous (IV) or subcutaneous (SC) infusion or an alternative treatment will be administered, as determined by the physician.
  Interventions: Biological: A licensed human normal immunoglobulin other than HYQVIA for IV or SC infusion or an alternative treatment
- HYQVIA Arm: Participant continues to receive HYQVIA (Immune Globulin (Human) 10% with recombinant human hyaluronidase (rHuPH20)), according to her treatment regimen.
  Interventions: Biological: HYQVIA [Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase]

INTERVENTIONS:
Biological: A licensed human normal immunoglobulin other than HYQVIA for IV or SC infusion or an alternative treatment — To be determined by the physician
  Groups: Alternative Product Arm
Biological: HYQVIA [Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase] — Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase
  Other Names: Hyqvia
  Groups: HYQVIA Arm

SUMMARY:
The purpose of this registry is to acquire safety data (including assessment of anti-rHuPH20 antibodies), regarding the course and outcome of pregnancy in women ever treated with HYQVIA. Development of the fetus/infant at birth and for the first 2 years will also be followed.

ELIGIBILITY:
Inclusion Criteria:

* For the expectant mother only: Participant became pregnant during or after treatment with HYQVIA
* Participant/Participant's legally authorized representative is willing to sign an informed consent form (ICF)

Exclusion Criteria:

* There are no applicable Exclusion Criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who became pregnant after ever treated with HYQVIA, and their infant children
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Director, Study Director — Shire
Locations (8):
- QuintilesIMS Plaza Building, Durham, North Carolina, United States
- Fakultni nemocnice Kralovske Vinohrady, Prague, Czechia
- Germany (3):
  - Freiburg University Hospital/ Prof. Dr. med. Bodo Grimbacher, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Klinikum St. Georg GmbH, Leipzig, Saxony
- Wojskowy Instytut Medyczny, Warsaw, Poland
- Slovakia (2):
  - Onkologicky ustav svatej Alzbety s.r.o., Bratislava
  - RAFMED s.r.o, Košice

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Borte M, Raffac S, Hrubisko M, Jahnz-Rozyk K, Garcia E, McCoy B, Chavan S, Nagy A, Yel L. Long-term safety of facilitated subcutaneous immunoglobulin treatment in pregnant women with primary immunodeficiency diseases: results from a registry study. Immunotherapy. 2022 Jun;14(8):609-616. doi: 10.2217/imt-2021-0336. Epub 2022 Apr 20. PMID 35443783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 centers in Czech Republic, Germany, Poland, Slovakia, and United States of America from 04 December 2015 (first participant first visit) to 17 December 2019 (last participant last visit).
Pre-assignment Details: Total 16 participants (9 mothers and 7 infants) were enrolled in the study. Of 9 mothers, 7 included in Retrospective (R) cohort and 2 in Prospective (P) cohort. Of 7 infants enrolled from 9 mothers (1 mother lost to follow-up; another mother withdrew consent prior to delivery) of R cohort; 5 included in R cohort and 2 included in P cohort. Study consisted of Study Arm1 (Alternative Product Arm) and Study Arm2 (HyQvia Arm). All participants were analyzed according to type of enrollment R and P.
Groups:
- Retrospective Cohort: Expectant Mothers: Participants (Expectant mothers) in the study arm 1 (Alternative Product arm) who stopped HYQVIA treatment (if the participant was still treated) and a licensed human normal immunoglobulin other than HYQVIA for intravenous (IV) or subcutaneous (SC) infusion or an alternative treatment were administered, as determined by the physician. Retrospective cohort included participants with condition of the fetus had been assessed through prenatal testing such as targeted ultrasound, via the antenatal diagnostic CRF, prior to the time of enrollment or the outcome of the pregnancy was known prior to the time of enrollment.
- Prospective Cohort: Expectant Mothers: Participants (Expectant mothers) in the study arm 2 (HyQvia Arm) continued to receive HYQVIA (Immune Globulin [Human] 10% with recombinant human hyaluronidase [rHuPH20]), according to her treatment regimen. Prospective cohort included participants with condition of the fetus had not been assessed through prenatal testing such as targeted ultrasound prior to the time of enrollment and the outcome of the pregnancy was not known at the time of enrollment.
- Retrospective Cohort: Infants: Participants (Infants) in the study arm 1 (Alternative Product arm) who stopped HYQVIA treatment (if the participant was still treated) and a licensed human normal immunoglobulin other than HYQVIA for IV or SC infusion or an alternative treatment were administered, as determined by the physician. Retrospective cohort included participants with condition of the fetus had been assessed through prenatal testing such as targeted ultrasound, via the antenatal diagnostic CRF, prior to the time of enrollment or the outcome of the pregnancy was known prior to the time of enrollment.
- Prospective Cohort: Infants: Participants (Infants) in the study arm 2 (HyQvia Arm) continued to receive HYQVIA (Immune Globulin [Human] 10% with recombinant human hyaluronidase [rHuPH20]), according to her treatment regimen. Prospective cohort included participants with condition of the fetus had not been assessed through prenatal testing such as targeted ultrasound prior to the time of enrollment and the outcome of the pregnancy was not known at the time of enrollment.
Period: Overall Study
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers | Retrospective Cohort: Infants | Prospective Cohort: Infants
Started | 7 | 2 | 5 | 2
Completed | 5 | 2 | 4 | 2
Not Completed | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Set consisted of all participants who had signed informed consent and meet all inclusion/exclusion criteria at the time of enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers | Retrospective Cohort: Infants | Prospective Cohort: Infants | Total
Number analyzed (Participants) | 7 | 2 | 5 | 2 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 5 | 2 | 7
  Between 18 and 65 years | 7 | 2 | 0 | 0 | 9
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 2 | 2 | 13
  Male | 0 | 0 | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 1 | 5 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 2 | 5 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a participant administered a medicinal product that did not necessarily had a causal relationship with the treatment. A SAE was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, is an important medical event. Number of participants with SAEs in expectant mothers and infants were reported.
Time Frame: From start of study drug administration up to end of study (up to 48.4 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers | Retrospective Cohort: Infants | Prospective Cohort: Infants
Number analyzed (Participants) | 7 | 2 | 5 | 2
Participants | 0 | 1 | 1 | 1

2. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs), Related and Not Related to HyQvia/Human Normal Immunoglobulin (IG) or Alternative Treatment
Description: An AE was defined as any untoward medical occurrence in a participant administered a medicinal product that did not necessarily have a causal relationship with the treatment. Number of participants with Non-SAEs, related and not related to HyQvia/Human Normal IG or alternative treatment in expectant mothers and infants were reported.
Time Frame: From start of study drug administration up to end of study (up to 48.4 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers | Retrospective Cohort: Infants | Prospective Cohort: Infants
Number analyzed (Participants) | 7 | 2 | 5 | 2
Participants
  Participants with Non-SAEs | 2 | 2 | 4 | 1
  Participants with AE related to human normal immunoglobulin treatment | 0 | 0 | 0 | 0
  Participants with AE related to HyQvia | 0 | 0 | 0 | 0
  Participants with AE related to alternative treatment | 0 | 0 | 0 | 0
  Participants: AE not related to HyQvia/human normal immunoglobulin treatment/alternative treatment | 2 | 2 | 4 | 2

3. Secondary Outcome: Number of Participants With Adverse Event of Special Interests (AESIs) in Expectant Mothers
Description: AESI were AEs that were considered by the sponsor to be relevant for the monitoring of the safety profile. AESI's included in this study were local/immunologic AEs including skin changes (Such as, local erythema, local pruritus, induration, nodules). Number of participants with AESIs in expectant mother were reported.
Time Frame: From start of first mother enrollment up to last mother's completion/discontinuation of study (up to 29.1 months)
Population: Enrolled set consisted of all participants who had signed informed consent and meet all inclusion/exclusion criteria at the time of enrollment. Data for this outcome was not planned to be collected and analyzed for infant group.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers
Number analyzed (Participants) | 7 | 2
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Who Developed Anti-rHuPH20 Antibodies in Expectant Mothers
Description: Number of participants who developed positive [titer ≥160] of anti-rHuPH20 binding in expectant mothers were reported. Neutralizing antibodies were assessed if the binding antibody assay has a result of 160 or above.
Time Frame: From start of first mother enrollment up to last mother's completion/discontinuation of study (up to 29.1 months)
Population: Enrolled set consisted of all participants who had signed informed consent and meet all inclusion/exclusion criteria at the time of enrollment. Data for this outcome was not planned to be collected and analyzed for infant group. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers
Number analyzed (Participants) | 3 | 1
Participants
  Anti-rHuPH20 binding antibody : Positive | 0 | 0
  Anti-rHuPH20 neutralizing antibody: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Antenatal Diagnostic Procedures
Description: Antenatal diagnostic procedures included ultrasound, serology and nuchal translucency screen which are used to assess the Fetal growth/development. Number of participants reported fetal growth/development were recorded.
Time Frame: Throughout the expectant mother pregnancy duration (up to 40 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers
Number analyzed (Participants) | 7 | 2
Participants
  Ultrasound | 3 | 0
  Serology | 2 | 0
  Nuchal Translucency Screen | 1 | 0

6. Secondary Outcome: Number of Participants Who Experienced General Pregnancy Outcomes
Description: Pregnancy outcomes included live birth, fetal death, termination or unknown.
Time Frame: Throughout the expectant mother pregnancy duration (up to 40 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers
Number analyzed (Participants) | 7 | 2
Participants
  Live Birth | 6 | 2
  Fetal Death | 0 | 0
  Termination | 0 | 0
  Missing | 1 | 0

7. Secondary Outcome: Number of Participants With Neonatal Assessment
Description: Neonatal assessment included parameters like weight, length, head circumference, Apgar scores, pulse rate, blood pressure, respiratory rate, body temperature with normal, abnormal and missing status. The Apgar scores was determined by evaluating the newborn baby on five simple criteria: Appearance, Pulse, Grimace, Activity, Respiration: on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Zero is the worst possible score and 10 is the highest possible score.
Time Frame: At or after delivery/end of pregnancy (up to 40 weeks)
Population: Enrolled set consisted of all participants who had signed informed consent and meet all inclusion/exclusion criteria at the time of enrollment. Data for this outcome was not planned to be collected and analyzed for Expectant mothers.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Infants | Prospective Cohort: Infants
Number analyzed (Participants) | 5 | 2
Participants
  Weight: Normal | 5 | 2
  Weight: Abnormal | 0 | 0
  Weight: Missing | 0 | 0
  Length: Normal | 5 | 1
  Length: Abnormal | 0 | 0
  Length: Missing | 0 | 1
  Head circumference: Normal | 4 | 0
  Head circumference: Abnormal | 0 | 0
  Head circumference: Missing | 1 | 2
  Apgar scores: Normal | 5 | 2
  Apgar scores: Abnormal | 0 | 0
  Apgar scores: Missing | 0 | 0
  Pulse rate: Normal | 0 | 0
  Pulse rate: Abnormal | 0 | 0
  Pulse rate: Missing | 5 | 2
  Blood pressure: Normal | 0 | 0
  Blood pressure: Abnormal | 0 | 0
  Blood pressure: Missing | 5 | 2
  Respiratory rate: Normal | 0 | 0
  Respiratory rate: Abnormal | 0 | 0
  Respiratory rate: Missing | 5 | 2
  Body temperature: Normal | 0 | 0
  Body temperature: Abnormal | 0 | 0
  Body temperature: Missing | 5 | 2

8. Secondary Outcome: Number of Participants With Status of the Infant at Birth
Description: Status of the infant at birth included the following as: Any need for resuscitation of the infant, Admission in intensive care unit, Presence of congenital malformations/anomaly, Any other conditions noted at or around birth with status yes, no and unknown.
Time Frame: At or after delivery/end of pregnancy (up to 40 weeks)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Infants | Prospective Cohort: Infants
Number analyzed (Participants) | 5 | 2
Participants
  Any need for resuscitation of the infant: Yes | 0 | 0
  Any need for resuscitation of the infant: No | 5 | 2
  Any need for resuscitation of the infant: Unknown | 0 | 0
  Admission in intensive care unit: Yes | 0 | 0
  Admission in intensive care unit: No | 5 | 2
  Admission in intensive care unit: Unknown | 0 | 0
  Presence of congenital malformations/anomaly: Yes | 1 | 1
  Presence of congenital malformations/anomaly: No | 4 | 1
  Presence of congenital malformations/anomaly: Unknown | 0 | 0
  Any other conditions noted at or around birth: Yes | 0 | 0
  Any other conditions noted at or around birth: No | 5 | 2
  Any other conditions noted at or around birth: Unknown | 0 | 0

9. Secondary Outcome: Number of Participants With Growth Measurement and Charts for the Infant
Description: Growth measurement and charts for the infant was assessed based on following parameters: Any congenital malformations diagnosed that were not reported at birth, any conditions that were noted since birth, weight assessment, length assessment, head circumference assessment. Number of participants with growth measurement and charts for the infant at 6, 12, 18 and 24 months follow-up was reported.
Time Frame: At 6, 12, 18 and 24 months follow-up
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Infants | Prospective Cohort: Infants
Number analyzed (Participants) | 5 | 2
Participants
  6 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Yes | 0 | 0
  6 months follow-up: Any congenital malformations diagnosed that were not reported at birth: No | 1 | 1
  6 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Unknown | 0 | 0
  6 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Missing | 4 | 1
  6 months follow-up: Any conditions that were noted since birth: Yes | 0 | 0
  6 months follow-up: Any conditions that were noted since birth: No | 1 | 1
  6 months follow-up: Any conditions that were noted since birth: Unknown | 0 | 0
  6 months follow-up: Any conditions that were noted since birth: Missing | 4 | 1
  6 months follow-up: Weight assessment: Normal | 1 | 2
  6 months follow-up: Weight assessment: Abnormal and clinically significant | 0 | 0
  6 months follow-up: Weight assessment: Abnormal but not clinically significant | 0 | 0
  6 months follow-up: Weight assessment: Missing | 4 | 0
  6 months follow-up: Length assessment: Normal | 1 | 1
  6 months follow-up: Length assessment: Abnormal and clinically significant | 0 | 0
  6 months follow-up: Length assessment: Abnormal but not clinically significant | 0 | 0
  6 months follow-up: Length assessment: Missing | 4 | 1
  6 months follow-up: Head circumference assessment: Normal | 1 | 1
  6 months follow-up: Head circumference assessment: Abnormal and clinically significant | 0 | 0
  6 months follow-up: Head circumference assessment: Abnormal but not clinically significant | 0 | 0
  6 months follow-up: Head circumference assessment: Missing | 4 | 1
  12 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Yes | 0 | 0
  12 months follow-up: Any congenital malformations diagnosed that were not reported at birth: No | 0 | 1
  12 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Unknown | 0 | 0
  12 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Missing | 5 | 1
  12 months follow-up: Any conditions that were noted since birth: Yes | 0 | 0
  12 months follow-up: Any conditions that were noted since birth: No | 0 | 1
  12 months follow-up: Any conditions that were noted since birth: Unknown | 0 | 0
  12 months follow-up: Any conditions that were noted since birth: Missing | 5 | 1
  12 months follow-up: Weight assessment: Normal | 1 | 1
  12 months follow-up: Weight assessment: Abnormal and clinically significant | 0 | 0
  12 months follow-up: Weight assessment: Abnormal but not clinically significant | 0 | 0
  12 months follow-up: Weight assessment: Missing | 4 | 1
  12 months follow-up: Length assessment: Normal | 1 | 1
  12 months follow-up: Length assessment: Abnormal and clinically significant | 0 | 0
  12 months follow-up: Length assessment: Abnormal but not clinically significant | 0 | 0
  12 months follow-up: Length assessment: Missing | 4 | 1
  12 months follow-up: Head circumference assessment: Normal | 1 | 1
  12 months follow-up: Head circumference assessment: Abnormal and clinically significant | 0 | 0
  12 months follow-up: Head circumference assessment: Abnormal but not clinically significant | 0 | 0
  12 months follow-up: Head circumference assessment: Missing | 4 | 1
  18 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Yes | 0 | 0
  18 months follow-up: Any congenital malformations diagnosed that were not reported at birth: No | 1 | 0
  18 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Unknown | 0 | 0
  18 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Missing | 4 | 2
  18 months follow-up: Any conditions that were noted since birth: Yes | 1 | 0
  18 months follow-up: Any conditions that were noted since birth: No | 0 | 0
  18 months follow-up: Any conditions that were noted since birth: Unknown | 0 | 0
  18 months follow-up: Any conditions that were noted since birth: Missing | 4 | 2
  18 months follow-up: Weight assessment: Normal | 1 | 0
  18 months follow-up: Weight assessment: Abnormal and clinically significant | 0 | 0
  18 months follow-up: Weight assessment: Abnormal but not clinically significant | 0 | 0
  18 months follow-up: Weight assessment: Missing | 4 | 2
  18 months follow-up: Length assessment: Normal | 1 | 0
  18 months follow-up: Length assessment: Abnormal and clinically significant | 0 | 0
  18 months follow-up: Length assessment: Abnormal but not clinically significant | 0 | 0
  18 months follow-up: Length assessment: Missing | 4 | 2
  18 months follow-up: Head circumference assessment: Normal | 1 | 0
  18 months follow-up: Head circumference assessment: Abnormal and clinically significant | 0 | 0
  18 months follow-up: Head circumference assessment: Abnormal but not clinically significant | 0 | 0
  18 months follow-up: Head circumference assessment: Missing | 4 | 2
  24 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Yes | 0 | 0
  24 months follow-up: Any congenital malformations diagnosed that were not reported at birth: No | 1 | 1
  24 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Unknown | 0 | 0
  24 months follow-up: Any congenital malformations diagnosed that were not reported at birth: Missing | 4 | 1
  24 months follow-up: Any conditions that were noted since birth: Yes | 0 | 0
  24 months follow-up: Any conditions that were noted since birth: No | 1 | 1
  24 months follow-up: Any conditions that were noted since birth: Unknown | 0 | 0
  24 months follow-up: Any conditions that were noted since birth: Missing | 4 | 1
  24 months follow-up: Weight assessment: Normal | 0 | 1
  24 months follow-up: Weight assessment: Abnormal and clinically significant | 0 | 0
  24 months follow-up: Weight assessment: Abnormal but not clinically significant | 0 | 0
  24 months follow-up: Weight assessment: Missing | 5 | 1
  24 months follow-up: Length assessment: Normal | 0 | 1
  24 months follow-up: Length assessment: Abnormal and clinically significant | 0 | 0
  24 months follow-up: Length assessment: Abnormal but not clinically significant | 0 | 0
  24 months follow-up: Length assessment: Missing | 5 | 1
  24 months follow-up: Head circumference assessment: Normal | 0 | 1
  24 months follow-up: Head circumference assessment: Abnormal and clinically significant | 0 | 0
  24 months follow-up: Head circumference assessment: Abnormal but not clinically significant | 0 | 0
  24 months follow-up: Head circumference assessment: Missing | 5 | 1

10. Secondary Outcome: Number of Participants With Development Milestones
Description: Developmental milestones evaluation included rolled over, attended to and reached for objects, sat up without support, turned to locate a voice, said his/her first words, and stand without support/help. Number of participants with development milestones at 6, 12, 18 and 24 months follow-up was reported.
Time Frame: At 6, 12, 18 and 24 months follow-up
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Cohort: Infants | Prospective Cohort: Infants
Number analyzed (Participants) | 5 | 2
Participants
  6 months follow-up: Rolled over: Not applicable yet | 0 | 0
  6 months follow-up: Rolled over: Milestone reached | 1 | 1
  6 months follow-up: Rolled over: Milestone missed | 0 | 0
  6 months follow-up: Rolled over: Unknown | 0 | 0
  6 months follow-up: Rolled over: Missing | 4 | 1
  6 months follow-up: Attended to and reached for objects: Not applicable yet | 0 | 0
  6 months follow-up: Attended to and reached for objects: Milestone reached | 1 | 1
  6 months follow-up: Attended to and reached for objects: Milestone missed | 0 | 0
  6 months follow-up: Attended to and reached for objects: Unknown | 0 | 0
  6 months follow-up: Attended to and reached for objects: Missing | 4 | 1
  6 months follow-up: Sat up without support: Not applicable yet | 1 | 0
  6 months follow-up: Sat up without support: Milestone reached | 0 | 1
  6 months follow-up: Sat up without support: Milestone missed | 0 | 0
  6 months follow-up: Sat up without support: Unknown | 0 | 0
  6 months follow-up: Sat up without support: Missing | 4 | 1
  6 months follow-up: Turned to locate a voice: Not applicable yet | 0 | 0
  6 months follow-up: Turned to locate a voice: Milestone reached | 1 | 1
  6 months follow-up: Turned to locate a voice: Milestone missed | 0 | 0
  6 months follow-up: Turned to locate a voice: Unknown | 0 | 0
  6 months follow-up: Turned to locate a voice: Missing | 4 | 1
  6 months follow-up: Said his/her first words: Not applicable yet | 1 | 1
  6 months follow-up: Said his/her first words: Milestone reached | 0 | 0
  6 months follow-up: Said his/her first words: Milestone missed | 0 | 0
  6 months follow-up: Said his/her first words: Unknown | 0 | 0
  6 months follow-up: Said his/her first words: Missing | 4 | 1
  6 months follow-up: Stand without support/help: Not applicable yet | 1 | 1
  6 months follow-up: Stand without support/help: Milestone reached | 0 | 0
  6 months follow-up: Stand without support/help: Milestone missed | 0 | 0
  6 months follow-up: Stand without support/help: Unknown | 0 | 0
  6 months follow-up: Stand without support/help: Missing | 4 | 1
  12 months follow-up: Rolled over: Not applicable yet | 0 | 0
  12 months follow-up: Rolled over: Milestone reached | 0 | 0
  12 months follow-up: Rolled over: Milestone missed | 0 | 0
  12 months follow-up: Rolled over: Unknown | 0 | 1
  12 months follow-up: Rolled over: Missing | 5 | 1
  12 months follow-up: Attended to and reached for objects: Not applicable yet | 0 | 0
  12 months follow-up: Attended to and reached for objects: Milestone reached | 0 | 0
  12 months follow-up: Attended to and reached for objects: Milestone missed | 0 | 0
  12 months follow-up: Attended to and reached for objects: Unknown | 0 | 1
  12 months follow-up: Attended to and reached for objects: Missing | 5 | 1
  12 months follow-up: Sat up without support: Not applicable yet | 0 | 0
  12 months follow-up: Sat up without support: Milestone reached | 0 | 0
  12 months follow-up: Sat up without support: Milestone missed | 0 | 0
  12 months follow-up: Sat up without support: Unknown | 0 | 1
  12 months follow-up: Sat up without support: Missing | 5 | 1
  12 months follow-up: Turned to locate a voice: Not applicable yet | 0 | 0
  12 months follow-up: Turned to locate a voice: Milestone reached | 0 | 0
  12 months follow-up: Turned to locate a voice: Milestone missed | 0 | 0
  12 months follow-up: Turned to locate a voice: Unknown | 0 | 1
  12 months follow-up: Turned to locate a voice: Missing | 5 | 1
  12 months follow-up: Said his/her first words: Not applicable yet | 0 | 0
  12 months follow-up: Said his/her first words: Milestone reached | 0 | 0
  12 months follow-up: Said his/her first words: Milestone missed | 0 | 0
  12 months follow-up: Said his/her first words: Unknown | 0 | 1
  12 months follow-up: Said his/her first words: Missing | 5 | 1
  12 months follow-up: Stand without support/help: Not applicable yet | 0 | 0
  12 months follow-up: Stand without support/help: Milestone reached | 0 | 0
  12 months follow-up: Stand without support/help: Milestone missed | 0 | 0
  12 months follow-up: Stand without support/help: Unknown | 0 | 0
  12 months follow-up: Stand without support/help: Missing | 5 | 2
  18 months follow-up: Rolled over: Not applicable ye | 0 | 0
  18 months follow-up: Rolled over: Milestone reached | 1 | 0
  18 months follow-up: Rolled over: Milestone missed | 0 | 0
  18 months follow-up: Rolled over: Unknown | 0 | 0
  18 months follow-up: Rolled over: Missing | 4 | 2
  18 months follow-up: Attended to and reached for objects: Not applicable yet | 0 | 0
  18 months follow-up: Attended to and reached for objects: Milestone reached | 1 | 0
  18 months follow-up: Attended to and reached for objects: Milestone missed | 0 | 0
  18 months follow-up: Attended to and reached for objects: Unknown | 0 | 0
  18 months follow-up: Attended to and reached for objects: Missing | 4 | 2
  18 months follow-up: Sat up without support: Not applicable yet | 0 | 0
  18 months follow-up: Sat up without support: Milestone reached | 1 | 0
  18 months follow-up: Sat up without support: Milestone missed | 0 | 0
  18 months follow-up: Sat up without support: Unknown | 0 | 0
  18 months follow-up: Sat up without support: Missing | 4 | 2
  18 months follow-up: Turned to locate a voice: Not applicable yet | 0 | 0
  18 months follow-up: Turned to locate a voice: Milestone reached | 1 | 0
  18 months follow-up: Turned to locate a voice: Milestone missed | 0 | 0
  18 months follow-up: Turned to locate a voice: Unknown | 0 | 0
  18 months follow-up: Turned to locate a voice: Missing | 4 | 2
  18 months follow-up: Said his/her first words: Not applicable yet | 0 | 0
  18 months follow-up: Said his/her first words: Milestone reached | 1 | 0
  18 months follow-up: Said his/her first words: Milestone missed | 0 | 0
  18 months follow-up: Said his/her first words: Unknown | 0 | 0
  18 months follow-up: Said his/her first words: Missing | 4 | 2
  18 months follow-up: Stand without support/help: Not applicable yet | 0 | 0
  18 months follow-up: Stand without support/help: Milestone reached | 1 | 0
  18 months follow-up: Stand without support/help: Milestone missed | 0 | 0
  18 months follow-up: Stand without support/help: Unknown | 0 | 0
  18 months follow-up: Stand without support/help: Missing | 4 | 2
  24 months follow-up: Rolled over: Not applicable yet | 0 | 0
  24 months follow-up: Rolled over: Milestone reached | 0 | 1
  24 months follow-up: Rolled over: Milestone missed | 0 | 0
  24 months follow-up: Rolled over: Unknown | 1 | 0
  24 months follow-up: Rolled over: Missing | 4 | 1
  24 months follow-up: Attended to and reached for objects: Not applicable yet | 0 | 0
  24 months follow-up: Attended to and reached for objects: Milestone reached | 0 | 1
  24 months follow-up: Attended to and reached for objects: Milestone missed | 0 | 0
  24 months follow-up: Attended to and reached for objects: Unknown | 1 | 0
  24 months follow-up: Attended to and reached for objects: Missing | 4 | 1
  24 months follow-up: Sat up without support: Not applicable yet | 0 | 0
  24 months follow-up: Sat up without support: Milestone reached | 1 | 1
  24 months follow-up: Sat up without support: Milestone missed | 0 | 0
  24 months follow-up: Sat up without support: Unknown | 0 | 0
  24 months follow-up: Sat up without support: Missing | 4 | 1
  24 months follow-up: Turned to locate a voice: Not applicable yet | 0 | 0
  24 months follow-up: Turned to locate a voice: Milestone reached | 1 | 1
  24 months follow-up: Turned to locate a voice: Milestone missed | 0 | 0
  24 months follow-up: Turned to locate a voice: Unknown | 0 | 0
  24 months follow-up: Turned to locate a voice: Missing | 4 | 1
  24 months follow-up: Said his/her first words: Not applicable yet | 0 | 0
  24 months follow-up: Said his/her first words: Milestone reached | 0 | 1
  24 months follow-up: Said his/her first words: Milestone missed | 0 | 0
  24 months follow-up: Said his/her first words: Unknown | 1 | 0
  24 months follow-up: Said his/her first words: Missing | 4 | 1
  24 months follow-up: Stand without support/help: Not applicable yet | 0 | 0
  24 months follow-up: Stand without support/help: Milestone reached | 1 | 1
  24 months follow-up: Stand without support/help: Milestone missed | 0 | 0
  24 months follow-up: Stand without support/help: Unknown | 0 | 0
  24 months follow-up: Stand without support/help: Missing | 4 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of study (up to 48.4 months)
Arm/Group | Retrospective Cohort: Expectant Mothers | Prospective Cohort: Expectant Mothers | Retrospective Cohort: Infants | Prospective Cohort: Infants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/2 | 1/5 | 1/2
Other Adverse Events (participants affected / at risk) | 2/7 | 2/2 | 4/5 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retrospective Cohort: Expectant Mothers (N=7) | Prospective Cohort: Expectant Mothers (N=2) | Retrospective Cohort: Infants (N=5) | Prospective Cohort: Infants (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cleft lip (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retrospective Cohort: Expectant Mothers (N=7) | Prospective Cohort: Expectant Mothers (N=2) | Retrospective Cohort: Infants (N=5) | Prospective Cohort: Infants (N=2)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02556775/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT02556775/SAP_001.pdf